CLINICAL TRIAL: NCT02956460
Title: Performance Comparison Between Fanfilcon A and Senofilcon A Sphere Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: EX-MKTG-73
Record Dates: First submitted 2016-11-03; First posted 2016-11-07 (Estimated); Results first posted 2017-12-08 (Actual); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- fanfilcon A (Active Comparator): Participants are randomized to wear fanfilcon A for two weeks during the cross over study.
  Interventions: Device: fanfilcon A
- senofilcon A (Active Comparator): Participants are randomized to wear senofilcon A for two weeks during the cross over study.
  Interventions: Device: senofilcon A

INTERVENTIONS:
Device: fanfilcon A — contact lens
  Arms: fanfilcon A
Device: senofilcon A — contact lens
  Arms: senofilcon A

SUMMARY:
Prospective, multi-center, bilateral, double-masked, randomized, cross-over, daily wear, 1 month dispensing study (2 weeks each lens pair)

DETAILED DESCRIPTION:
The aim of this study is to determine the clinical performance of fanfilcon A in comparison to senofilcon A sphere contact lenses.

ELIGIBILITY:
Inclusion Criteria:

A person is eligible for inclusion in the study if he/she:

* Is between 18 and 40 years of age (inclusive)
* Has read, understood and signed the information consent letter
* Has had a self-reported eye exam in the last two years
* Is a spherical soft contact lens wearer
* Has a contact lens prescription that fits within the available parameters of the study lenses
* Has a spectacle cylinder no greater than 0.75D (Diopters) in each eye
* Can achieve best corrected spectacle distance visual acuity of 20/25 (0.10 logMAR) or better in each eye
* Can achieve a distance visual acuity of 20/30 (0.18 logMAR) or better in each eye with the study contact lenses
* Has clear corneas and no active ocular disease
* Is willing and anticipated to be able to comply with the wear schedule (8 hours per day; 5 days a week of lens wear)
* Is willing and able to follow instructions and maintain the appointment schedule

Exclusion Criteria:

A person will be excluded from the study if he/she:

* Has a history of not achieving comfortable CL (Contact Lens) wear (defined as 5 days per week; >8 hours/day)
* Is currently wearing senofilcon C (2 weeks lens), senofilcon A 1-Day, senofilcon C (monthly lens) or enfilcon A contact lenses
* Is habitually using rewetting/ lubricating eye drops more than once per day
* Presents with clinically significant anterior segment abnormalities
* Presents with ocular or systemic disease or need of medications which might interfere with contact lens wear
* Presents with slit lamp findings that would contraindicate contact lens wear such as:

  * Pathological dry eye or associated findings
  * Significant pterygium, pinguecula, or corneal scars within the visual axis
  * Neovascularization > 0.75 mm in from of the limbus
  * Giant papillary conjunctivitis (GCP) worse than grade 1
  * Anterior uveitis or iritis (or history in past year)
  * Seborrheic eczema of eyelid region, Seborrheic conjunctivitis
  * History of corneal ulcers or fungal infections
  * Poor personal hygiene
* Has a known history of corneal hypoesthesia (reduced corneal sensitivity)
* Has aphakia, keratoconus or a highly irregular cornea
* Has presbyopia or has dependence on spectacles for near work over the contact lenses
* Has undergone corneal refractive surgery

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2016-10-27 (Actual); Primary Completion 2016-12-14 (Actual); Study Completion 2016-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Jones, PhD, FAAO, Study Director — Centre for Contact Lens Research
Locations (4):
- United States (4):
  - Eric M. White O. D., Inc, San Diego, California
  - Golden Vision, Sarasota, Florida
  - Kannarr Eye Care, Pittsburg, Kansas
  - Nittany Eye Associates, State College, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Fanfilcon A First Then Senofilcon A: Participants are randomized to wear fanfilcon A for two weeks then senofilcon A
- Senofilcon A First Then Fanfilcon A: Participants are randomized to wear senofilcon A for two weeks then fanfilcon A
Period: Lens 1
Arm/Group | Fanfilcon A First Then Senofilcon A | Senofilcon A First Then Fanfilcon A
Started | 30 | 34
Completed | 29 | 34
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Period: Lens 2
Arm/Group | Fanfilcon A First Then Senofilcon A | Senofilcon A First Then Fanfilcon A
Started | 29 | 34
Completed | 29 | 34
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fanfilcon A First Then Senofilcon A | Senofilcon A First Then Fanfilcon A | Total
Number analyzed (Participants) | 30 | 34 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.6 (6.1) | 29.6 (5.6) | 30.5 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 28 | 52
  Male | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Overall Comfort
Description: Subjective assessment for comfort is assessed. Scale 0-10, 0=painful, 10=can't feel
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Fanfilcon A: Participants are randomized to wear fanfilcon A either first or second for two weeks during the cross over study.
- Senofilcon A: Participants are randomized to wear senofilcon A either first or second for two weeks during the cross over study.
Arm/Group | Fanfilcon A | Senofilcon A
Number analyzed (Participants) | 63 | 63
units on a scale | 8.4 (1.9) | 8.7 (1.5)

2. Primary Outcome: Overall Dryness
Description: Subjective ratings for dryness is assessed on a scale of 0-10, 0=extremely dry, 10=no dryness
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fanfilcon A | Senofilcon A
Number analyzed (Participants) | 63 | 63
units on a scale | 8.2 (1.9) | 8.2 (1.9)

3. Primary Outcome: Vision Quality
Description: Subjective ratings of vision quality is assessed on a scale 0-10, 0=not sharp/not clear, 10=sharp/clear
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fanfilcon A | Senofilcon A
Number analyzed (Participants) | 63 | 63
units on a scale | 9.0 (1.5) | 8.9 (1.6)

4. Primary Outcome: Lens Handling
Description: Subjective ratings of lens handling - insertion and removal - is assessed using scale 0-10, 0=difficult to handle, 10=very easy to handle
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fanfilcon A | Senofilcon A
Number analyzed (Participants) | 63 | 63
units on a scale
  Insertion | 9.3 (1.3) | 9.4 (1.2)
  Removal | 8.4 (2.0) | 9.3 (1.3)

5. Primary Outcome: Vision Satisfaction
Description: Subjective ratings of vision satisfaction is assessed on a scale 0-10, 0=completely dissatisfied, 10=completely satisfied.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fanfilcon A | Senofilcon A
Number analyzed (Participants) | 63 | 63
units on a scale | 8.7 (2.1) | 8.6 (1.7)

6. Primary Outcome: Lens Centration
Description: Lens centration will be recorded by degree and direction in the primary position. (Optimum, decentration acceptable, decentration unacceptable).
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Fanfilcon A | Senofilcon A
Number analyzed (Participants) | 63 | 63
Participants
  Optimum | 62 | 63
  Acceptable | 1 | 0
  Unacceptable | 0 | 0

7. Primary Outcome: Conjunctival Staining
Description: Assessed using slit lamp with blue light and sodium fluorescein, low medium magnification.
  0=None, no staining present
  1. Very slight
  2. Slight
  3. Moderate
  4. Severe
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fanfilcon A | Senofilcon A
Number analyzed (Participants) | 63 | 63
units on a scale | 0.4 (0.7) | 0.6 (0.8)

8. Primary Outcome: Smoothness
Description: Subjective ratings for lens sensation of smoothness is assessed on a scale 0-10, 0=not smooth at all, 10=totally smooth
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fanfilcon A | Senofilcon A
Number analyzed (Participants) | 63 | 63
units on a scale | 8.7 (1.7) | 9.1 (1.4)

9. Primary Outcome: Clean Feeling
Description: Subjective ratings for lens clean feeling is assessed on a scale 0-10, 0=not clean at all, 10=lenses feel perfectly clean
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fanfilcon A | Senofilcon A
Number analyzed (Participants) | 63 | 63
units on a scale | 8.7 (1.7) | 8.9 (1.4)

10. Primary Outcome: Lens Hydrated
Description: Subjective ratings for lens sensation is assessed on a scale 0-10, 0=totally dehydrated, 10=totally hydrated
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fanfilcon A | Senofilcon A
Number analyzed (Participants) | 63 | 63
units on a scale | 8.3 (2.0) | 8.5 (1.6)

11. Primary Outcome: Lens Wettability
Description: Subjective ratings for lens wettability is assessed on a scale 0-10, 0=non-wettable, 10=highly wettable
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fanfilcon A | Senofilcon A
Number analyzed (Participants) | 63 | 63
units on a scale | 8.4 (1.9) | 8.5 (1.6)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the 2 week period for each lens
Arm/Group | Fanfilcon A | Senofilcon A
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/63
Other Adverse Events (participants affected / at risk) | 0/63 | 0/63

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure restriction on the PI is that the sponsor should be notified of any use of study data for results communication.